CLINICAL TRIAL: NCT05559476
Title: A Phase 3, Open-label, Randomized, Controlled, Multicountry Study to Evaluate the Immune Response, Safety and Reactogenicity of RSVPreF3 OA Investigational Vaccine When Co-administered With FLU HD Vaccine in Adults Aged 65 Years and Above
Brief Title: A Study on the Immune Response and Safety Elicited by a Vaccine Against Respiratory Syncytial Virus (RSV) When Given Alone and Together With a Vaccine Against Influenza in Adults Aged 65 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 214489; 2021-001356-34 (EudraCT Number)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; High dose quadrivalent influenza vaccine; Immunogenicity; Safety; Reactogenicity; Adults aged 65 years and above
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Co-Ad Group (Experimental): Participants received one dose of FLU-HD vaccine and one dose of RSVPreF3 OA vaccine, both doses administered at Day 1, and were followed until end of study.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: FLU HD vaccine
- Control Group (Active Comparator): Participants received one dose of FLU-HD vaccine at Day 1, followed by one dose of RSVPreF3 OA vaccine at Day 31, and were followed until the study end.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: FLU HD vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — RSVPreF3 OA investigational vaccine administered intramuscularly in the deltoid region of the non-dominant arm.
Biological: FLU HD vaccine — FLU HD vaccine administered intramuscularly in the deltoid region of the dominant arm (Co-Ad Group) or the non-dominant arm (Control Group).

SUMMARY:
The purpose of this study is to assess the immunogenicity, safety and reactogenicity of the RSVPreF3 OA investigational vaccine when co-administered with the high dose quadrivalent influenza (FLU HD) vaccine in adults aged 65 years and above compared to separate administration of the vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* A male or female ≥65 years of age at the time of the first study intervention administration.
* Participants living in the general community or in an assisted-living facility that provides minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Written or witnessed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Participants who are medically stable in the opinion of the investigator at the time of first vaccination. Participants with chronic stable medical conditions with or without specific treatment are allowed to participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Hypersensitivity to latex.
* History of Guillain Barré syndrome, or anaphylaxis.
* Serious or unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or un-controlled neurological disorders or seizures. Participants with medically-controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol (e.g. completion of diary cards, attend regular phone calls/study site visits).
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study interventions during the period beginning 30 days before the first study vaccine administration, or planned use during the study period.
* Administration of an influenza vaccine during the 6 months preceding the study FLU vaccine administration.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration.

Note: In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is recommended and/or organized by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.

* Previous vaccination with an RSV vaccine.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the first dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first study vaccination or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other exclusions

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Planned move during the study conduct that prohibits participation until 1 month post-last vaccine administration.
* Bedridden participants.
* Participation of any study personnel or their immediate dependents, family, or household members.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Canoga Park, California
  - GSK Investigational Site, Colton, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Immokalee, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Sandy Springs, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Mishawaka, Indiana
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Ames, Iowa
  - GSK Investigational Site, El Dorado, Kansas
  - GSK Investigational Site, Methuen, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, North Las Vegas, Nevada
  - GSK Investigational Site, Warren Township, New Jersey
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Rocky Mount, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Edmond, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Jefferson City, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Buynak R, Cannon K, DeAtkine D, Kirby J, Usdan L, Bhavsar A, Gerard C, Kuznetsova A, Jayadev A, Amare H, Valenciano S, Meyer N. Randomized, Open-Label Phase 3 Study Evaluating Immunogenicity, Safety, and Reactogenicity of RSVPreF3 OA Coadministered with FLU-QIV-HD in Adults Aged >/= 65. Infect Dis Ther. 2024 Aug;13(8):1789-1805. doi: 10.1007/s40121-024-00985-4. Epub 2024 Jun 26. PMID 38981954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1029 participants received at least one dose of the study intervention and were included in the exposed set.
Pre-assignment Details: This study assessed the immunogenicity, safety and reactogenicity of the RSVPre3 OA vaccine when co-administered with Flu High-Dose vaccine (FLU-HD [FLU]), in adults aged 65 years old or above.
Period: Overall Study
Arm/Group | Co-Ad Group | Control Group
Started | 516 | 513
Completed | 493 | 485
Not Completed | 23 | 28
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 13 | 12
Not completed — Consent withdrawal, not due to a (S)AE | 8 | 14
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-Ad Group | Control Group | Total
Number analyzed (Participants) | 516 | 513 | 1029
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 71.3 (5.3) | 71.1 (5.1) | 71.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 243 | 510
  Male | 249 | 270 | 519
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alasaka Native | 4 | 6 | 10
  Asian | 4 | 4 | 8
  Black or African American | 72 | 68 | 140
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 355 | 352 | 707
  Other, Not Specified | 81 | 82 | 163

OUTCOME MEASURES:

1. Primary Outcome: RSV-A Neutralizing Titers Expressed as Group Geometric Mean Titers (GMTs)
Description: RSV-A neutralizing titers were given as group GMTs and expressed as Estimated Dilution 60 (ED60).
Time Frame: At 1 month after the RSVPreF3 OA vaccine dose (Day 31 for the Co-Ad Group and Day 61 for the Control Group)
Population: Analysis was performed on Per Protocol Set (PPS) for RSV analysis which included eligible participants who: received RSVPreF3 OA vaccine dose in Control group and all study doses in Co-Ad group, had pre and post-dose immunogenicity results, adhered to specified blood draw intervals, had immunogenicity data available for the specified analysis at the specified time point post-RSVPreF3 OA vaccine dose, lacked interfering medical conditions and avoided prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 457 | 414
Titers | 5876.3 [5299.5 to 6515.9] | 6935.3 [6200.0 to 7757.9]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the RSVPreF3 OA vaccine when co-administered with the FLU vaccine compared to the RSVPreF3 OA vaccine administered alone, in terms of RSV-A neutralizing antibody titers, at 1 month after the RSVPreF3 OA vaccine dose (Day 31 for the Co-Ad Group and Day 61 for the Control Group); Test type: Non-Inferiority — The non-inferiority is demonstrated if the Upper Limit (UL) of the 2-sided 95% Confidence Interval (CI) of the GMT ratio (Control group divided by Co-Ad group) for RSVPreF3 OA vaccine is less than or equal (<=)1.5; GMT Ratio = 1.18, 95% CI 2-sided [1.03 to 1.35] — The comparison is done using the adjusted group ratio of GMT (ANCOVA model applied to the logarithm- transformed titers). The ANCOVA model included the treatment group, the age category as fixed effects and the pre-dose log-10 titer as covariate

2. Primary Outcome: Hemagglutinin Inhibition (HI) Titers for 4 FLU Vaccine Strains Expressed as Group GMTs
Description: HI titers were assessed against the Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata strains.
Time Frame: At 1 month after the FLU vaccine dose (Day 31 for both groups)
Population: Analysis was performed on PPS for FLU analysis which included eligible participants who: received FLU vaccine dose in Control group and all study doses in Co-Ad group, had pre- and post-dose immunogenicity results, adhered to specified blood draw intervals, had immunogenicity data available for the specified analysis at the specified time point post-FLU vaccine dose, lacked interfering medical conditions and avoided prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 456 | 440
Titers
  Flu A/Darwin/6/2021 H3N2 | 72.7 [64.1 to 82.5] | 72.3 [63.7 to 82.1]
  Flu A/Victoria/2570/2019 H1N1: number analyzed (Participants) | 450 | 434
  Flu A/Victoria/2570/2019 H1N1 | 189.9 [167.6 to 215.1] | 177.3 [156.4 to 200.9]
  Flu B/Austria/1359417/2021 Victoria | 859.8 [805.8 to 917.5] | 820.9 [768.8 to 876.6]
  Flu B/Phuket/3073/2013 Yamagata: number analyzed (Participants) | 454 | 440
  Flu B/Phuket/3073/2013 Yamagata | 758.7 [699.1 to 823.4] | 703.4 [647.7 to 763.9]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone, in terms of HI GMTs against the Flu A/Darwin/6/2021 H3N2 influenza strain, at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI of the group GMT ratio (Control group divided by Co-Ad group) for HI antibody titers for the Flu strain is <=1.5; GMT Ratio = 0.99, 95% CI 2-sided [0.85 to 1.16] — The comparison was done using the adjusted group ratio of GMT (ANCOVA model applied to the logarithm- transformed titers). The ANCOVA model included the treatment group, the age category as fixed effects and the pre-dose log-10 titer as covariate
Statistical Analysis 2: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone, in terms of HI GMTs against the Flu A/Victoria/2570/2019 H1N1 influenza strain, at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMT Ratio = 0.93, 95% CI 2-sided [0.80 to 1.09] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the FLU vaccine when co administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone, in terms of HI GMTs against the Flu B/Austria/1359417/2021 influenza strain, at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMT Ratio = 0.95, 95% CI 2-sided [0.88 to 1.03] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the FLU vaccine when co administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone, in terms of HI GMTs against the Flu B/Phuket/3073/2013 Yamagata influenza strain, at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMT Ratio = 0.93, 95% CI 2-sided [0.84 to 1.02] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: RSV-B Neutralizing Titers Expressed as Group GMTs
Description: RSV-B neutralizing titers were given as group GMTs and expressed as Estimated Dilution 60 (ED60).
Time Frame: At 1 month after the RSVPreF3 OA vaccine dose (Day 31 for the Co-Ad Group and Day 61 for the Control Group)
Population: Analysis was performed on PPS for RSV analysis which included eligible participants who: received RSVPreF3 OA vaccine dose in Control group and all study doses in Co-Ad group, had pre- and post-dose immunogenicity results, adhered to specified blood draw intervals, had immunogenicity data available for the specified analysis at the specified time point post- RSVPreF3 OA vaccine dose, lacked interfering medical conditions and avoided prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 457 | 355
Titers | 8251.5 [7460.6 to 9126.3] | 8359.0 [7492.8 to 9325.3]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the RSVPreF3 OA vaccine when co-administered with the FLU vaccine compared to the RSVPreF3 OA vaccine administered alone, in terms of RSV-B neutralizing antibody titers, at 1 month after the RSVPreF3 OA vaccine dose (Day 31 for the Co-Ad Group and Day 61 for the Control Group); Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI of the GMT ratio (Control group divided by Co-Ad group) for RSVPreF3 OA vaccine is <=1.5; GMT Ratio = 1.01, 95% CI 2-sided [0.89 to 1.15] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: HI Seroconversion Rate (SCR) for 4 FLU Vaccine Strains
Description: SCR for HI titers was defined as the percentage of participants who have either a HI predose titer less than (<) 1:10 and a post-dose titer greater than or equal to (>=) 1:40, or a pre-dose titer >= 1:10 and at least a 4-fold increase in post-dose titer. The assessed Flu strains were: Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata.
Time Frame: At 1 month after the FLU vaccine dose (Day 31 for both groups)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 456 | 440
Percentage of participants
  Flu A/Darwin/6/2021 H3N2 | 59.2 [54.5 to 63.8] | 57.5 [52.7 to 62.2]
  Flu A/Victoria/2570/2019 H1N1: number analyzed (Participants) | 450 | 434
  Flu A/Victoria/2570/2019 H1N1 | 50.9 [46.2 to 55.6] | 46.8 [42.0 to 51.6]
  Flu B/Austria/1359417/2021 Victoria | 39.7 [35.2 to 44.3] | 31.1 [26.8 to 35.7]
  Flu B/Phuket/3073/2013 Yamagata: number analyzed (Participants) | 454 | 440
  Flu B/Phuket/3073/2013 Yamagata | 43.6 [39.0 to 48.3] | 37.7 [33.2 to 42.4]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To evaluate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone as measured by the difference of percentage of participants achieving seroconversion for HI antibody titers against Flu A/Darwin/6/2021 H3N2 strain at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI on the group difference (Control group minus Co-Ad group) in terms of SCR is <=10% for anti-HI antibodies; Difference of Percentage = -1.71, 95% CI 2-sided [-8.15 to 4.74]
Statistical Analysis 2: Comparison: Co-Ad Group vs Control Group; To evaluate the non-inferiority of the FLU vaccine when co administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone as measured by the difference of percentage of participants achieving seroconversion for HI antibody titers against Flu A/Victoria/2570/2019 H1N1 strain at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Difference of Percentage = -4.11, 95% CI 2-sided [-10.67 to 2.48]
Statistical Analysis 3: Comparison: Co-Ad Group vs Control Group; To evaluate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone as measured by the difference of percentage of participants achieving seroconversion for HI antibody titers against Flu B/Austria/1359417/2021 Victoria at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Difference of Percentage = -8.56, 95% CI 2-sided [-14.75 to -2.29]
Statistical Analysis 4: Comparison: Co-Ad Group vs Control Group; To evaluate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone as measured by the difference of percentage of participants achieving seroconversion for HI antibody titers against Flu B/Phuket/3073/2013 Yamagata strain at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Difference of Percentage = -5.89, 95% CI 2-sided [-12.28 to 0.56]

5. Secondary Outcome: RSV-A Neutralizing Titers Expressed as Mean Geometric Increase (MGI)
Description: MGI was defined as the geometric mean of the within-participant ratios of the post-dose titer over the pre-dose titer.
Time Frame: At 1 month after the RSVPreF3 OA vaccine dose (Day 31 for the Co-Ad Group and Day 61 for the Control Group) compared to pre-vaccination (Day 1 for Co-Ad group and Day 31 for Control group)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 457 | 356
Ratio | 5.59 [5.02 to 6.23] | 6.75 [5.93 to 7.68]

6. Secondary Outcome: RSV-B Neutralizing Titers Expressed as MGI
Description: MGI was defined as the geometric mean of the within-participant ratios of the post-dose titer over the pre-dose titer.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 457 | 355
Ratio | 5.19 [4.69 to 5.75] | 5.29 [4.65 to 6.03]

7. Secondary Outcome: HI Titers for Each of the 4 FLU Vaccine Strains Expressed as GMT
Description: HI titers were assessed against the Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata strains. HI antibodies were expressed as GMTs, in titers.
Time Frame: At Day 1 and 1 month after FLU vaccine dose administration (Day 31 for both groups)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 507 | 503
Titers
  Flu A/Darwin/6/2021 H3N2, Day 1 | 11.5 [10.5 to 12.7] | 12.6 [11.4 to 14.0]
  Flu A/Darwin/6/2021 H3N2, Day 31: number analyzed (Participants) | 457 | 440
  Flu A/Darwin/6/2021 H3N2, Day 31 | 71.8 [63.6 to 81.0] | 75.1 [66.7 to 84.4]
  Flu A/Victoria/2570/2019 H1N1, Day 1: number analyzed (Participants) | 500 | 495
  Flu A/Victoria/2570/2019 H1N1, Day 1 | 35.3 [31.2 to 40.1] | 41.9 [36.9 to 47.6]
  Flu A/Victoria/2570/2019 H1N1, Day 31: number analyzed (Participants) | 455 | 440
  Flu A/Victoria/2570/2019 H1N1, Day 31 | 200.0 [178.7 to 223.8] | 194.7 [173.9 to 217.9]
  Flu B/Austria/1359417/2021 Victoria, Day 1 | 292.6 [270.6 to 316.4] | 308.5 [285.8 to 333.1]
  Flu B/Austria/1359417/2021 Victoria, Day 31: number analyzed (Participants) | 457 | 440
  Flu B/Austria/1359417/2021 Victoria, Day 31 | 848.0 [799.7 to 899.2] | 818.3 [769.2 to 870.5]
  Flu B/Phuket/3073/2013 Yamagata, Day 1: number analyzed (Participants) | 505 | 503
  Flu B/Phuket/3073/2013 Yamagata, Day 1 | 239.2 [220.6 to 259.3] | 245.5 [226.1 to 266.5]
  Flu B/Phuket/3073/2013 Yamagata, Day 31: number analyzed (Participants) | 457 | 440
  Flu B/Phuket/3073/2013 Yamagata, Day 31 | 751.1 [698.9 to 807.2] | 699.6 [646.9 to 756.6]

8. Secondary Outcome: HI Seroprotection Rate (SPR) for 4 FLU Vaccine Strains
Description: SPR for HI titers was defined as the percentage of participants with a serum HI titer >= 1:40. The assessed Flu strains were: The assessed Flu strains were: Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata.
Time Frame: At Day 1 and 1 month after FLU vaccine dose administration (Day 31 for both groups)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 507 | 503
Percentage of participants
  Flu A/Darwin/6/2021 H3N2, Day 1 | 17.9 [14.7 to 21.6] | 21.9 [18.3 to 25.7]
  Flu A/Darwin/6/2021 H3N2, Day 31: number analyzed (Participants) | 457 | 440
  Flu A/Darwin/6/2021 H3N2, Day 31 | 75.3 [71.1 to 79.2] | 76.6 [72.3 to 80.5]
  Flu A/Victoria/2570/2019 H1N1, Day 1: number analyzed (Participants) | 500 | 495
  Flu A/Victoria/2570/2019 H1N1, Day 1 | 53.4 [48.9 to 57.8] | 61.0 [56.6 to 65.3]
  Flu A/Victoria/2570/2019 H1N1, Day 31: number analyzed (Participants) | 455 | 440
  Flu A/Victoria/2570/2019 H1N1, Day 31 | 92.3 [89.5 to 94.6] | 94.5 [92.0 to 96.5]
  Flu B/Austria/1359417/2021 Victoria, Day 1 | 98.8 [97.4 to 99.6] | 99.6 [98.6 to 100.0]
  Flu B/Austria/1359417/2021 Victoria, Day 31: number analyzed (Participants) | 457 | 440
  Flu B/Austria/1359417/2021 Victoria, Day 31 | 100 [99.2 to 100] | 100 [99.2 to 100]
  Flu B/Phuket/3073/2013 Yamagata, Day 1: number analyzed (Participants) | 505 | 503
  Flu B/Phuket/3073/2013 Yamagata, Day 1 | 96.8 [94.9 to 98.2] | 98.2 [96.6 to 99.2]
  Flu B/Phuket/3073/2013 Yamagata, Day 31: number analyzed (Participants) | 457 | 440
  Flu B/Phuket/3073/2013 Yamagata, Day 31 | 100 [99.2 to 100] | 100 [99.2 to 100]

9. Secondary Outcome: HI Titers for 4 FLU Vaccine Strains, Expressed as MGI
Description: MGI was defined as the geometric mean of the within-participant ratios of the post-dose titer over the pre-dose titer.
Time Frame: At 1 month after the FLU vaccine dose administration (Day 31 for both groups)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 456 | 440
Ratio
  Flu A/Darwin/6/2021 H3N2 | 6.20 [5.49 to 7.00] | 5.87 [5.20 to 6.62]
  Flu A/Victoria/2570/2019 H1N1: number analyzed (Participants) | 450 | 434
  Flu A/Victoria/2570/2019 H1N1 | 5.57 [4.81 to 6.46] | 4.53 [3.94 to 5.21]
  Flu B/Austria/1359417/2021 Victoria | 2.92 [2.69 to 3.18] | 2.71 [2.51 to 2.93]
  Flu B/Phuket/3073/2013 Yamagata: number analyzed (Participants) | 454 | 440
  Flu B/Phuket/3073/2013 Yamagata | 3.13 [2.85 to 3.44] | 2.87 [2.62 to 3.14]

10. Secondary Outcome: Percentage of Participants With Solicited Administration Site Events After Each Vaccine Dose Administration
Description: The solicited administration site events after vaccination included erythema, pain and swelling.
Time Frame: Within 4 days (the day of vaccination and 3 subsequent days) after each vaccination (administered on Day 1 and 31)
Population: Analysis was performed on Modified Safety Set, which included participants who received a study intervention, with the electronic diary completed post-each vaccination by the participant or authorized caregiver, and for whom solicited administration event data was available for the specific visit. The Control group received FLU vaccination at Day 1 and RSVPreF3 OA vaccination at Day 31; Co-Ad group received co-administered vaccine (RSVPreF3 OA + FLU) on Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 423 | 414
Percentage of participants
  Erythema, Flu administration at Day 1 | 4.0 [2.4 to 6.4] | 4.6 [2.8 to 7.1]
  Erythema, RSV administration at Day 1: number analyzed (Participants) | 423 | 0
  Erythema, RSV administration at Day 1 | 4.3 [2.5 to 6.6] |
  Erythema, RSV administration at Day 31: number analyzed (Participants) | 0 | 400
  Erythema, RSV administration at Day 31 |  | 4.3 [2.5 to 6.7]
  Pain, Flu administration at Day 1 | 47.0 [42.2 to 51.9] | 43.5 [37.7 to 47.4]
  Pain, RSV administration at Day 1: number analyzed (Participants) | 423 | 0
  Pain, RSV administration at Day 1 | 55.6 [50.7 to 60.4] |
  Pain, RSV administration at Day 31: number analyzed (Participants) | 0 | 400
  Pain, RSV administration at Day 31 |  | 45.8 [40.8 to 50.8]
  Swelling, Flu administration at Day 1 | 4.5 [2.7 to 6.9] | 5.6 [3.6 to 8.2]
  Swelling, RSV administration at Day 1: number analyzed (Participants) | 423 | 0
  Swelling, RSV administration at Day 1 | 4.0 [2.4 to 6.4] |
  Swelling, RSV administration at Day 31: number analyzed (Participants) | 0 | 400
  Swelling, RSV administration at Day 31 |  | 4.3 [2.5 to 6.7]

11. Secondary Outcome: Percentage of Participants Reporting Each Solicited Systemic Event After Each Vaccine Dose Administration
Description: The solicited systemic events after vaccination include arthralgia, fatigue, fever, headache and myalgia.
Time Frame: Within 4 days (the day of vaccination and 3 subsequent days) after each vaccination (administered on Day 1 and 31)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 423 | 493
Percentage of participants
  Arthralgia, Dosing at Day 1: number analyzed (Participants) | 423 | 414
  Arthralgia, Dosing at Day 1 | 16.1 [12.7 to 19.9] | 13.8 [10.6 to 15.5]
  Arthralgia, Dosing at Day 31: number analyzed (Participants) | 0 | 400
  Arthralgia, Dosing at Day 31 |  | 13.0 [9.9 to 16.7]
  Fatigue, Dosing at Day 1: number analyzed (Participants) | 423 | 414
  Fatigue, Dosing at Day 1 | 30.5 [26.1 to 35.1] | 22.0 [18.1 to 26.3]
  Fatigue, Dosing at Day 31: number analyzed (Participants) | 0 | 400
  Fatigue, Dosing at Day 31 |  | 23.5 [19.4 to 28.0]
  Fever, Dosing at Day 1: number analyzed (Participants) | 423 | 424
  Fever, Dosing at Day 1 | 2.1 [1.0 to 4.0] | 0.7 [0.1 to 2.1]
  Fever, Dosing at Day 31: number analyzed (Participants) | 0 | 400
  Fever, Dosing at Day 31 |  | 2.0 [0.9 to 3.9]
  Headache, Dosing at Day 1: number analyzed (Participants) | 423 | 414
  Headache, Dosing at Day 1 | 24.3 [20.3 to 28.7] | 17.1 [13.6 to 21.1]
  Headache, Dosing at Day 31: number analyzed (Participants) | 0 | 400
  Headache, Dosing at Day 31 |  | 19.0 [15.3 to 23.2]
  Myalgia, Dosing at Day 1: number analyzed (Participants) | 423 | 414
  Myalgia, Dosing at Day 1 | 40.2 [35.5 to 45.0] | 34.1 [29.5 to 38.8]
  Myalgia, Dosing at Day 31: number analyzed (Participants) | 0 | 400
  Myalgia, Dosing at Day 31 |  | 31.3 [26.7 to 36.0]

12. Secondary Outcome: Percentage of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited AEs is an AE that is not included in a list of solicited events using a participant diary. Unsolicited events must have been spontaneously communicated by a participant who signs the informed consent. Unsolicited AEs include both serious, non-serious AEs and potential immune-mediated diseases (pIMDs).
Time Frame: Within 30 days after vaccine administration (the day of vaccination and 29 subsequent days after vaccination)
Population: Analysis was performed on Exposed set which included participants who received a study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 516 | 513
Percentage of participants | 12.2 [9.5 to 15.3] | 13.5 [10.6 to 16.7]

13. Secondary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant.
Time Frame: From Day 1 up to study end (6 months after last vaccination - Month 6 for Co-Ad Group and Month 7 for Control group)
Population: Analysis was performed on Exposed set which included participants who received a study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 516 | 513
Percentage of participants | 2.3 [1.2 to 4.0] | 2.9 [1.6 to 4.8]

14. Secondary Outcome: Percentage of Participants Reporting Potential Immune-mediated Disease (pIMDs)
Description: pIMDs are a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. The investigator must exercise his/her medical/scientific judgment to determine whether other diseases have an autoimmune origin (i.e. pathophysiology involving systemic or organ-specific pathogenic autoantibodies) and should also be recorded as a pIMD.
Time Frame: From Day 1 up to study end (6 months after last vaccination - Month 6 for Co-Ad Group and Month 7 for Control group)
Population: Analysis was performed on Exposed set which included participants who received a study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 516 | 513
Percentage of participants | 0 [0 to 0.7] | 0.4 [0.0 to 1.4]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during 4-day follow-up period after each vaccination. Unsolicited AEs were collected during 30-day follow-up period after each vaccination. SAEs and pIMDs were collected throughout the study period (from Day 1 to study end [6 months after last vaccination]).
Description: Solicited and unsolicited events were reported per participant at any dose for the assessed timeframe (within 30 days after any vaccine dose administration) according to occurence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | Co-Ad Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/516 | 0/513
Serious Adverse Events (participants affected / at risk) | 12/516 | 15/513
Other Adverse Events (participants affected / at risk) | 339/516 | 319/513
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=516) | Control Group (N=513)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Spinal cord infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=516) | Control Group (N=513)
Injection site pain (General disorders) | 273 (274) | 257 (371)
Fatigue (General disorders) | 130 (132) | 140 (185)
Injection site swelling (General disorders) | 27 (27) | 34 (40)
Pyrexia (General disorders) | 11 (11) | 13 (13)
Chills (General disorders) | 0 (0) | 4 (4)
Injection site pruritus (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 2 (2) | 2 (2)
Administration site erythema (General disorders) | 1 (1) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 1 (1)
Administration site pruritus (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site paraesthesia (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 73 (73) | 91 (109)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 113 (115) | 128 (157)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (6)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 4 (4) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 4 (5)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale acute (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 27 (27) | 34 (40)
Myalgia (Musculoskeletal and connective tissue disorders) | 177 (177) | 203 (270)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT05559476/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT05559476/SAP_001.pdf